CLINICAL TRIAL: NCT00456833
Title: A Combined Phase 1 and 2 Study Investigating the Combination of RAD001 and Erlotinib in Patients With Advanced NSCLC Previously Treated Only With Chemotherapy
Brief Title: Combination of RAD001 and Erlotinib in Patients With Advanced Non Small Cell Lung Cancer Previously Treated Only With Chemotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C2111; 2004-003017-16 (EudraCT Number)
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2012-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC; Advanced lung cancer; RAD; RAD001; erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Everolimus; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAD 5mg/day + erlotinib (Experimental)
  Interventions: Drug: RAD001
- erlotinib 150mg/day (Active Comparator)
  Interventions: Drug: RAD001; Drug: erlotinib

INTERVENTIONS:
Drug: RAD001
Drug: erlotinib
  Arms: erlotinib 150mg/day

SUMMARY:
This study aims to assess the value of combined treatment with RAD001 and erlotinib in patients with advanced Non Small Cell Lung Cancer treated only with chemotherapy as systemic therapy.

ELIGIBILITY:
Inclusion criteria:

* Age over 18 years
* Advanced Non Small Cell Lung Cancer which is not responding to chemotherapy treatment including either cisplatin or carboplatin
* Only 1-2 previous chemotherapy regimens for advanced disease
* More than 2 weeks from previous surgery, radiation or chemotherapy
* Ability to perform normal daily functions

Exclusion criteria:

* Chronic steroid treatment
* Prior treatment with EGFR inhibitors
* Active bleeding conditions, skin conditions, gastrointestinal disorders, mouth ulcers, eye conditions or other severe medical conditions
* Other cancers within the past 2 years
* Pregnant or breastfeeding women Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2005-06; Primary Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Phase 1: Dose limiting toxicities (DLT) and PK drug-drug interaction (DDI) measured during first 28 days of combined treatment for each treatment regimen and dose. | first 28 days of combined treatment
Phase 2: Tumor response assessed by CT scans measured at baseline and after 8 weeks of treatment for each feasible dose/regimen determined in phase 1 | at baseline and after 8 weeks of treatment

SECONDARY OUTCOMES:
Phase 1: Tumor response assessed by CT scans measured at baseline, monthly until month 4 then q2months until progression | at baseline, monthly until month 4 then q2months until progression
Phase 2: Safety and steady state drug levels evaluated monthly | Monthly
Phase 1 and 2: Exploratory Biomarker assessment from archival tumor tissue | Dec 2009

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (14):
- United States (7):
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Rochester, Minnesota
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Madison, Wisconsin
- Canada (3):
  - Novartis Investigative Site, Richmond, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Herlev, Denmark
- France (2):
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Villejuif
- Novartis Investigative Site, Moscow, Russia

REFERENCES:
- See also: Results for CRAD001C2111 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5703